CLINICAL TRIAL: NCT05931796
Title: Enhanced Recovery vs Conventional Recovery After Anesthesia for Patients Undergoing Breast Surgery
Brief Title: Enhanced vs Conventional Recovery After Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amal Gouda Elsayed Safan (Other)
Collaborators: Mahmoud Saeed Ebaid (Unknown)
Responsible Party: Sponsor-Investigator, Amal Gouda Elsayed Safan, lecturer of anaethesia, Menoufia University
Organization: Menoufia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3/2023ANET45
Record Dates: First submitted 2023-06-02; First posted 2023-07-05 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): NON-ERAS pathway All patients received best of care practice, with standardization of preoperative and postoperative care
  Interventions: Other: NON-ERAS pathway
- Group B (Active Comparator): ERAS pathway ERAS consist of approximately 15 elements (or components) that include preoperative, intraoperative, and postoperative interventions .
  Interventions: Other: ERAS pathway

INTERVENTIONS:
Other: NON-ERAS pathway — All patients received best of care practice, with standardization of preoperative and postoperative care
  Arms: Group A
Other: ERAS pathway — ERAS pathway ERAS consist of approximately 15 elements (or components) that include preoperative, intraoperative, and postoperative interventions .
  Arms: Group B

SUMMARY:
the investigators hypothesize that with the use of enhanced recovery of surgery (ERAS), the postoperative hospital stay after breast surgeries is reduced and also postoperative complications are decreased.

DETAILED DESCRIPTION:
Group A NON-ERAS pathway All patients received best of care practice, with standardization of preoperative and postoperative care. Group B ERAS pathway

ELIGIBILITY:
Inclusion Criteria:

* • Age: 20-60 years.

  * Adequate cognitive state (able to understand and collaborate)
  * American society of anesthesia (ASA) I, II

Exclusion Criteria:

* Patients who are:

  * Uncooperative.
  * Having allergy to any of the study drugs.
  * Known abuse of alcohol or medication.
  * Having Local infection at the site of injection or systemic infection.
  * Pregnancy.
  * With coagulation disorders.
  * Any complicated patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
This study aims to explore the effectiveness and safety of the enhanced recovery after surgery (ERAS) protocol vs. traditional perioperative care programs for modified radical mastectomy. | 48 hours
  visual analogue scale VAS Score (a scale from 0 to 10 where 0 is interpreted as no pain, 1- 4 mild pain, 5-6 moderate pain, 7-10 severe pain) will be recorded 15 min after extubation (as soon as the patient will be alert enough to report pain)' every 1hour for the first 8hours' then every 3hours for the remaining 24 hours.

SECONDARY OUTCOMES:
Time of first ambulation | 48 hours
  hours

OTHER OUTCOMES:
Anesthesia recovery time | hour
  minutes
Time to regular diet. | 24 hours
  hours
Postoperative opioid use. | 48h
  mg

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Saeed Ebaid, Principal Investigator — Menoufia University
Locations (1):
- Menoufia university, Cairo, Shibin Elkom, Egypt

IPD SHARING:
Plan to Share IPD: No